CLINICAL TRIAL: NCT00644293
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Three-Day Azithromycin for the Treatment of Group A β-Hemolytic Streptococcal Pharyngitis/Tonsillitis in Adolescents and Adults
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin Sustained Release Versus 3-Day Azithromycin for the Treatment of Strep Throat in Adolescents and Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661119
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Pharyngitis; Tonsillitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: azithromycin (Zithromax); Drug: placebo
- 2 (Experimental)
  Interventions: Drug: azithromycin SR; Drug: placebo

INTERVENTIONS:
Drug: azithromycin (Zithromax) — azithromycin 500 mg tablet by mouth once daily for 3 days
  Arms: 1
Drug: placebo — placebo
  Arms: 1
Drug: azithromycin SR — azithromycin SR 2.0 g by mouth as an oral slurry for 1 dose
  Arms: 2
Drug: placebo — placebo
  Arms: 2

SUMMARY:
To determine if a single 2.0-g dose of azithromycin SR is at least as effective as a 3-day course of azithromycin (500 mg once daily for 3 days) when used to treat adolescents and adults with strep throat, and to assess efficacy and safety for both treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of acute group A beta-hemolytic streptococcus (GABHS) pharyngitis/tonsillitis and a positive rapid antigen detection test or positive culture of the pharynx or tonsils for GABHS

Exclusion Criteria:

* Patients were excluded if they had treatment with any systemic antibiotic within the previous 7 days, a history of rheumatic fever, a peritonsillar abcess, or were known carriers of GABHS.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2003-01; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
bacteriologic response in the Bacteriologic per Protocol population | Test of Cure (TOC) visit (Days 24-28)

SECONDARY OUTCOMES:
sponsor assessment of clinical response in the Bacteriologic per Protocol population | TOC visit
bacteriologic response for the remaining study populations | TOC visit
sponsor assessment of clinical response for the Bacteriologic per Protocol population | Long-Term Follow-Up (LTFU) visit (Days 38-45)
bacteriologic response for the Bacteriologic per Protocol population | TOC visit
summary of baseline susceptibilities | Study endpoint
adverse events | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- United States (11):
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Nampa, Idaho
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Bensalem, Pennsylvania
  - Pfizer Investigational Site, Harleysville, Pennsylvania
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, West Jordan, Utah
- Belgium (3):
  - Pfizer Investigational Site, Erembodegem
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Hasselt
- Finland (2):
  - Pfizer Investigational Site, Nokia
  - Pfizer Investigational Site, Tampere
- France (6):
  - Pfizer Investigational Site, Courbevoie
  - Pfizer Investigational Site, Gentilly
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Villejuif
- Germany (7):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Erkner
  - Pfizer Investigational Site, Ludwigshafen
  - Pfizer Investigational Site, Rüdersdorf
  - Pfizer Investigational Site, Tostedt
  - Pfizer Investigational Site, Villingen-Schwenningen
  - Pfizer Investigational Site, Würzburg
- India (4):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Hyderabad
  - Pfizer Investigational Site, Pune
- Italy (5):
  - Pfizer Investigational Site, Foligno, PG
  - Pfizer Investigational Site, Gualdo Tadino, PG
  - Pfizer Investigational Site, S.Eraclio-Foligno, PG
  - Pfizer Investigational Site, Spoleto, PG
  - Pfizer Investigational Site, Vocabolo Gaifana-Gualdo Tadino, PG
- Netherlands (3):
  - Pfizer Investigational Site, Ede (Gld)
  - Pfizer Investigational Site, Geldermalsen
  - Pfizer Investigational Site, Huizen
- Norway (2):
  - Pfizer Investigational Site, Elverum
  - Pfizer Investigational Site, Skedsmokorset
- United Kingdom (8):
  - Pfizer Investigational Site, Bath, Avon
  - Pfizer Investigational Site, Hastings, East Sussex
  - Pfizer Investigational Site, Glenrothes, Fife
  - Pfizer Investigational Site, High Valleyfield, Fife
  - Pfizer Investigational Site, Tunbrige Wells, Kent
  - Pfizer Investigational Site, Atherstone, Warwickshire
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Kent

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661119&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Comparative%20Trial%20of%20Azithromycin%20Sustained%20Release%20Versus%203-Day%20Azithromycin%20for%20th